CLINICAL TRIAL: NCT02913196
Title: A Phase I Trial of Apalutamide Plus Abiraterone Acetate, Docetaxel, and Prednisone in Patients With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Phase I Trial of Apalutamide Plus Abiraterone Acetate, Docetaxel, and Prednisone in Patients With mCRPC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1509016578
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — apalutamide; Abiraterone Acetate; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Apalutamide, 120 mg (cohort 1), 240 mg (cohort 2), 180 mg (cohort 3) Abiraterone Acetate 1000mg Prednisone 10mg Docetaxel 75 mg/m2
  Interventions: Drug: Apalutamide; Drug: Abiraterone acetate; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Apalutamide — Orally available, small molecule, nonsteroidal potent and selective antagonist of the androgen receptor.
  Cohort 1 dose: 120 mg QD Cohort 2 dose: 240 mg QD Cohort 3 dose: 180 mg QD
  Other Names: ARN-509
Drug: Abiraterone acetate — Abiraterone acetate is the prodrug of the active drug abiraterone. Once absorbed after oral administration, abiraterone acetate is rapidly converted to the active form, abiraterone.
  Dose: 1000 mg QD
  Other Names: Zytiga
Drug: Docetaxel — Taxane cytotoxic chemotherapy with demonstrated survival benefit in those with advanced prostate cancer.
  Dose: 75 mg/m2 Q3W
  Other Names: Taxotere
Drug: Prednisone — Dose: 5 mg BID
  Other Names: Deltasone

SUMMARY:
This is a multi-center, Phase I study of apalutamide in combination with abiraterone acetate, docetaxel and prednisone in patients with metastatic mastrate resistant prostate cancer (mCRPC).

This study is designed to determine the dose that apalutamide can be administered safely in combination with abiraterone acetate, docetaxel and prednisone.

DETAILED DESCRIPTION:
Subjects are enrolled in up to three 3-6-subject cohorts and are administered combination (apalutamide, abiraterone acetate and docetaxel plus prednisone) according to a dose-escalation schedule. The first dose of docetaxel infusion begins on Day 1 Cycle 1. Daily oral apalutamide, abiraterone acetate plus twice-daily oral prednisone begins on Day 1 Cycle 1. Docetaxel 1-hour infusions are administered intravenously every 3 weeks (Q3W), preceded by oral dexamethasone. While a subject is receiving chemotherapy, a treatment cycle is defined as 21 days. Dose limiting toxicity (DLT) determination is based on toxicities observed within the initial 2 cycles defined as 6 weeks. DLT will be assessed before the start of the third docetaxel infusion. Once a combination dose is determined to be safe (i.e. no more than 2 of 6 subjects experience DLT), the next cohort will enroll. Subjects remain at their allocated combination dose until the maximum tolerated dose (MTD) is determined.

The primary objective is to determine a safe dose combination of apalutamide plus abiraterone acetate, docetaxel, prednisone in subjects with mCRPC.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on at least one of the following criteria:

   1. PSA progression according to Prostate Cancer Working Group 3 (PCWG3) criteria
   2. Objective radiographic progression in soft tissue, according to modified Response Evaluation Criteria In Solid Tumors (RECIST) or bone scans
3. ECOG performance status of 0-2
4. Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone orchiectomy
5. Age >18 years
6. Patients must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count >1,500/cells/mm3
   2. Hemoglobin ≥ 9 g/dL
   3. Platelet count >100,000 x 109/microliter
   4. Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault
   5. Serum albumin ≥3.2 g/dL
   6. Serum potassium ≥3.5 mmol/L
7. Patients must be able to take oral medication without crushing, dissolving or chewing tablets
8. Ability to understand and the willingness to sign a written informed consent document
9. Medications known to lower the seizure threshold (see list under prohibited medications) must be discontinued or substituted at least 4 weeks prior to study drug initiation
10. Patients on stable dose of bisphosphonates or RANK-L inhibitor, Denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication

Exclusion Criteria

1. Liver Function

   1. If total bilirubin is >1.5 x ULN (NOTE: in subjects with Gilbert's syndrome, if total bilirubin is >1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is within normal range, subject may be eligible) or
   2. Alanine (ALT) or aspartate (AST) aminotransferase >1.5xULN (or >5xULN for subject with liver metastasis) concomitant with alkaline phosphatase >2.5xULN (or >5xULN for subjects with bone or liver metastases) or
   3. Alanine (ALT or aspartate (AST) aminotransferase >2.5xULN (or >5xULN for subjects with liver metastasis
2. Use of investigational drugs (including vaccines) or implantation of invasive medical device ≤4 weeks or <5 half-lives of Cycle 1, Day 1 or current enrollment in investigational drug or device study
3. Prior exposure to apalutamide. Prior exposure to abiraterone acetate and/or other CYP17 inhibitors, enzalutamide is allowed (but not preferred) only during the dose escalation period
4. Prior chemotherapy for advanced prostate cancer. Prior chemotherapy for any other disease within 3 years
5. Prior systemic beta-emitting bone-seeking radioisotopes (i.e. strontium-90)
6. Pre-existing neuropathy ≥Grade 2
7. Systemic azole treatment (e.g. Fluconazole, itracanozole) ≤2 weeks of Cycle 1 Day 1
8. Use of potent inducers or inhibitors of CYP3A4 activity ≤2 weeks prior to Day 1 Cycle 1
9. History of adrenal insufficiency or hyperaldosteronism
10. Active or symptomatic viral hepatitis
11. Chronic liver disease
12. Brain metastases or leptomeningeal disease
13. Known allergies, hypersensitivity or intolerance to abiraterone acetate, apalutamide, docetaxel, dexamethasone, prednisone, or their excipients
14. Use of herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc) must be discontinued before treatment start. Daily Multi-vitamin, calcium and Vitamin D is allowed
15. Surgery or local prostatic intervention within 30 days of first dose. [Note: Any clinically relevant sequelae from surgery must have resolved prior to Day 1 Cycle 1]
16. Radiation therapy for treatment of prostate cancer ≤4 weeks of Day 1 Cycle 1
17. Current evidence of any of the following:

    1. Uncontrolled hypertension (defined as blood pressure of >150 mmHg systolic and/or >100 mmHg diastolic on medication)
    2. Gastrointestinal disorder affecting absorption
    3. Active infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
    4. Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily
    5. Any condition that in the opinion of the investigator, would preclude participation in this study
    6. Patients with baseline severe hepatic impairment (Child Pugh Class C)
18. Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to treatment start or New York Heart Association (NYHA) Class II to IV heart disease
19. Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
20. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 week after last study drug administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLT) | From the time of study drug administration till PSA progression or study completion (~36 months)
  Dose limiting toxicities will be measured by using the Common Terminology Criteria for Adverse Events or CTCAE version 4.0 which uses a grading scale from 1-5.

SECONDARY OUTCOMES:
Change in the number of subjects with prostate-specific antigen (PSA) response | Starting after 12 weeks, at the beginning of Week 4 of combination therapy with docetaxel, apalutamide, abiraterone acetate plus prednisone until PSA progression or study completion (~36 months)
Change in PSA response | At the start of treatment until PSA progression or study completion (~36 months)
  PSA response will be captured through blood sample collection and radiographic scans
Change in the time to PSA progression | At the start of treatment until PSA progression or study completion (~36 months)
  PSA progression will be determined by protocol-specific/modified Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
Change is radiographic progression-free survival | Images will be collected at baseline, 12 weeks and at end of study, an average of 100 months
  Radiographic progression will be determined via scans metric of CT, MRI and Bone scans
Change in CellSearch circulating tumor cells (CTC) enumration | Collected at baseline, 12 weeks and at end of study, an average of 100 months
  CTCs will be collected via blood sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Ana Molina, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No